CLINICAL TRIAL: NCT00351988
Title: Effects of Cancer Symptoms on Minority Caregivers
Brief Title: Effects of Cancer Symptoms on Caregivers
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2005-0404; 5 KO7 CA 102482-02 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Psychosocial
Keywords: Lung Cancer; Non-Small Cell Lung Cancer; Breast Cancer; Psychosocial; Behavioral; Caregiver; Interview; Questionnaire; Minority Caregiver; Non-Minority Caregiver; Survey
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- African American caregivers: African American caregivers for patients with advanced non-small cell lung cancer or breast cancer.
  Interventions: Behavioral: Phenomenological Interviews; Behavioral: Quantitative Interviews
- Latino caregivers: Latino caregivers for patients with advanced non-small cell lung cancer or breast cancer.
  Interventions: Behavioral: Phenomenological Interviews; Behavioral: Quantitative Interviews
- White non-Latino caregivers: White non-Latino caregivers for patients with advanced non-small cell lung cancer or breast cancer.
  Interventions: Behavioral: Phenomenological Interviews; Behavioral: Quantitative Interviews

INTERVENTIONS:
Behavioral: Phenomenological Interviews — Part 1 will collect phenomenologic data to understand the meaning of caregiver burden, and the positive experiences faced when caring for a underserved patient with advanced lung cancer.
Behavioral: Quantitative Interviews — Part 2 will collect quantitative data to determine the prevalence and severity of symptoms experienced by caregivers and their contribution to caregiver burden.
  Other Names: Questionnaire

SUMMARY:
The primary objectives are to:

1.1 identify and compare the experiences of minority and nonminority caregivers, including the prevalence and severity of physical (fatigue, sleep disturbance) and psychologic (depression, anxiety, stress) symptoms and their influence on caregiver symptom burden; and to

1.2 assess the relationship between caregiver's symptoms (physical and psychologic) and the patient's symptom's at multiple time points over the patient's treatment regimen for advanced solid tumors (lung, breast, cervical, and others).

A secondary objective is to:

1.3 describe the experience of being a minority (African American/Black or Latino) or nonminority person caring for a medically underserved patient with advanced solids tumors (lung, breast, cervical, or others) over the course of the patient's treatment regimen and follow-up clinic visits.

DETAILED DESCRIPTION:
Caregiver:

If you choose to take part in this study, you will be asked to complete 3 study visits over a period of about 20 weeks (the first visit, followed by 2 more visits, usually 3-8 weeks apart). During the first and third visits, you will be asked to take part in an interview that will include questions about your experience as a caregiver to a patient with cancer. The interview will last about 30-45 minutes and will be tape recorded. The text of the interviews will be copied from the tapes to a written format. The study staff will review the content to look for key caregiver concerns and experiences. The PI and study staff will be the only ones who will have access to the tapes and transcripts. All tapes will be destroyed after the study is finished.

You will also be asked to complete some brief surveys about your physical and psychological health, your reactions to being a caregiver, and your beliefs about symptoms and their control. It will take about 30-45 minutes to complete the surveys, each time.

Each study visit will take about 60-90 minutes. If you can not come to the clinic, trained research study staff will contact you by telephone or by a home visit (with your permission) to complete the surveys and interview. After the last of the 3 study visits, your participation will be ended in this study.

This is an investigational study. Up to 125 participants will take part in this multicenter study at 4 sites: Lyndon Baines Johnson Hospital, Ben Taub General Hospital, MD Anderson, and locations in the community identified by the participant and the study team. Up to 40 will be enrolled at MD Anderson.

Patient:

If you choose to take part in this study, you will be asked to complete 3 study visits over a period of about 20 weeks (the first visit, followed by 2 more visits, usually 3-8 weeks apart). During the visits, you will also be asked to complete some surveys about your physical and psychological health, your reactions to your caregiver, and your beliefs about symptoms and their control. It will take about 30 minutes to complete the surveys each time.

Each study visit will take about 45 minutes. If you can not come to the clinic, trained research study staff will contact you by telephone or by a home visit (with your permission) to complete the surveys and interview. After the last of the 3 study visits, your participation in this study will end.

This is an investigational study. Up to 125 patients will take part in this multicenter study at 4 sites: Lyndon Baines Johnson Hospital, Ben Taub General Hospital, MD Anderson and locations in the community identified by the participant and study team. Up to 40 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Caregiver inclusion criteria includes: provides care and/or assistance to a patient receiving new or current treatment - Single or combined chemotherapy, radiotherapy, and/or targeted therapy for advanced solid tumors (lung, breast, cervical, and other).
2. 18 years of age or older;
3. self-identified as African-American/Black, Latino, or white, non-Latino;
4. able to speak English or Spanish (as applicable);
5. able to read and complete forms or be willing to have the forms read to them by a trained interviewer;
6. accessible through personal or telephone contact for the duration of the study.
7. Patient inclusion criteria: Receiving new or current treatment - Single or combined - chemotherapy, radiotherapy, and/or targeted therapy for advanced solid tumors (lung, breast, cervical, and others). Criteria 2-6 are the same as listed under Caregiver Criteria.

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three groups of caregivers: African American, Latinos, and white non-Latinos.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2006-01-26 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Difference in reduction in psychological (depression, anxiety, stress) and physical symptoms (fatigue, sleep disturbance) between 3 groups of caregivers: African American, Latinos, and white non-Latinos | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Palos, DrPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Jackson Memorial, Miami, Florida
  - Lyndon Baines Johnson Hospital, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org